CLINICAL TRIAL: NCT05283460
Title: The Effect of Mandala Activity on Life Satisfaction of Women Receiving Chemotherapy for Gynecological Cancer: A Randomized Controlled Study
Brief Title: The Effect of Mandala Activity on Life Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Munzur University (Other)
Responsible Party: Principal Investigator, Nursel Alp Dal, Principal Investigator, Munzur University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: munzur u
Record Dates: First submitted 2022-02-07; First posted 2022-03-17 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: ART; Life Satisfaction; Gynecologic Cancer
Keywords: Gynecologic Cancer; Life satisfaction; Mandala
MeSH Terms: conditions — Personal Satisfaction | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This study was designed as a randomized controlled prospective double-blind clinical trial.
Who Masked: Participant, Care Provider
Masking Description: participants will not known wich type of group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mandala (Experimental): As in the case of previous studies, to prevent confusion and make the mandala drawing process easier, a few videos describing what a mandala is were shown to the patients, and information was provided. Next, each patient was given a set of felt-tip pens (in 24 different colors) and ready-to-use mandala papers, and they were asked to complete the mandala activity. The patients were given empty mandala books with enough pages for them to draw mandalas every day, they were asked to perform the mandala activity regularly in a time interval of their own choice every day, and whether they performed the activity was checked daily without them noticing (so that they would not have the feeling of being checked on or inspected).
  Interventions: Behavioral: mandala
- control group (No Intervention): The Life Satisfaction Scale was administered to patients in the control group at the first encounter (pre-test) and three weeks after the first encounter (post-test). Although the pre- and post-test treatment protocols were the same for both intervention and control groups, the only difference between their treament was the mandala activity, which was not applied to those in the control group. Patients in the control group continued their routine lives at home for three weeks. After the application, the mandala activity was applied to all patients who wanted it.

INTERVENTIONS:
Behavioral: mandala — The Life Satisfaction Scale was administered to patients in the control group at the first encounter (pre-test) and three weeks after the first encounter (post-test). Although the pre- and post-test treatment protocols were the same for both intervention and control groups, the only difference between their treament was the mandala activity, which was not applied to those in the control group. Patients in the control group continued their routine lives at home for three weeks. After the application, the mandala activity was applied to all patients who wanted it.
  Other Names: control group
  Arms: mandala

SUMMARY:
This study aimed to determine the effect of mandala activity on life satisfaction of women receiving chemotherapy for gynecological cancer.

DETAILED DESCRIPTION:
Data will be collected using the descriptive information form and the Life Satisfaction Scale.

ELIGIBILITY:
Inclusion Criteria:

* Receiving chemotherapy
* No communication problems
* Having at least 6 months of cancer diagnosis
* Being in Stage 2 and Stage 3 of the disease

Exclusion Criteria:

* Having a medical device (IV catheter, etc.) or physical symptoms (vision problems, Parkinson's disease, etc.) that may prevent mandala drawing.
* Being in Stage 1 and Stage 4 of the disease.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Because gynecological cancers occur only in women
Enrollment: 60 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Life satisfaction scale mean | up to 3 weeks
  Average score from life satisfaction scale ( Minimum score; 5, Maximum score;25)

SECONDARY OUTCOMES:
Life satisfaction scale mean | through study completion, an average of 1 year
  Average score from life satisfaction scale( Minimum score;5 , Maximum score;25)

CONTACTS AND LOCATIONS:
Overall Officials: Nursel A Dal, Assist Prof, Principal Investigator — Munzur Ünivesitesi
Locations (1):
- Munzur University, Tunceli, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No